CLINICAL TRIAL: NCT00300664
Title: A Randomized Trial of Human Growth Hormone (hGH) vs Placebo in Intensively Treated Haemato-Oncology Patients.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2128
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-03

CONDITIONS: Multiple Myeloma; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Multiple Myeloma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Human Growth Hormone

INTERVENTIONS:
Drug: Human Growth hormone

SUMMARY:
About 90% of patients with haemato-oncologic malignancy lose their body muscle mass and also lose weight either due to chemotherapy induced nausea/vomiting or the high catabolic state due to fever, sepsis or chemotherapy. This impacts tremendously on the days in hospital and also on the treatment-related complications. Studies with Human Growth hormone (hGH) have shown that it increases lean body mass in adult patients with AIDS and animal models of cancer. At the same time, in vitro studies have shown that hGH has no effect on tumor cell growth. This study is designed to see if the use of hGH in immunocompromised patients with haematological malignancies prevents the loss of muscle mass and weight loss to some extent.

This will be a blinded 1:1, randomised study including 150 patients whereby the patients will either receive hGH or a placebo. The doctors and the nurses will not know what drug the patient is receiving. Both hGH and the placebo will be given intravenously (if patients are receiving other intravenous antibiotics or haemopoietic support ) or subcutaneously (if platelets are above 20 x 109/L) The treatment will start on the first day of treatment and continue for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

- Age >= 18 years 2. Patients with haematological malignancies receiving neutropenia (< 0.5 x 109/L) inducing chemotherapy (+/- TBI) requiring hospitalisation.

3. Negative pregnancy test if the patient is of childbearing potential 4. Informed consent

Exclusion Criteria:

* . Previous treatment with growth hormone 2.Unstable psychiatric conditions 3. Uncontrolled endocrine disorders 4.Chronic severe liver disease: AST or ALT>3x upper limit of normal range 5. Chronic severe renal disease: creatinine>150 µM or repeated positive test for haematuria or proteinuria 6. Severe congestive heart failure 7. Aortic stenosis associated with clinical symptoms eg syncope of angina pectoris 8. Hypertrophic cardiomyopathy 9. Uncontrolled hypertension (diastolic blood-pressure > 105 mm Hg) 10. Diabetes mellitus that is not well controlled with insulin/antidiabetic drugs 11. Severe respiratory disease 12. Known or suspected allergy to growth hormone or any of its constituents 13. History of drug or alcohol abuse within two years prior to study enrolment 14. Exposure to another investigational medication or device currently or within three months prior to enrolment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-07; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Ray Powles, FRCP, FRCPath, Principal Investigator — Royal Marsden NHS Foundation Trust